CLINICAL TRIAL: NCT04472104
Title: Mindfulness-based Treatment for Sexual Difficulties Following Breast Cancer
Brief Title: BREast Cancer And Sexuality Treatment
Acronym: BREAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Lori Brotto, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H19-02480
Record Dates: First submitted 2019-11-19; First posted 2020-07-15 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-05

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: 3-year, randomized, unblinded, two-site, controlled trial of 8 weekly sessions of group Mindfulness-Based Cognitive Therapy for sexuality (MBCT-S) vs. 8 weekly sessions of a sex education treatment.
Who Masked: Outcomes Assessor
Masking Description: Those doing data analysis are blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBCT-S (Active Comparator): Mindfulness-Based Cognitive Therapy for sexuality (MBCT-S) which incorporates several empirically supported therapeutic approaches, integrating elements of education, mindfulness meditation skills, and sex therapy.
  Interventions: Behavioral: MBCT-S
- SexEd (Active Comparator): Sexuality education on sexual desire, sexual distress, and sexual pain.
  Interventions: Behavioral: SexEd

INTERVENTIONS:
Behavioral: MBCT-S — Group mindfulness treatment for sexual desire, sexual distress, and sexual pain in breast cancer (BrCa) survivors.
  Arms: MBCT-S
Behavioral: SexEd — Group sex education on sexual desire, sexual distress, and sexual pain in breast cancer (BrCa) survivors.
  Arms: SexEd

SUMMARY:
The purpose of this project is to compare the effects of a group mindfulness treatment versus a group sex education on sexual desire, sexual distress, and sexual pain in breast cancer (BrCa) survivors. Participants will be randomly assigned to either 8 weekly sessions of a group mindfulness-based treatment or 8 weekly sessions of a sex education group. Groups will consist of approximately 8 breast cancer survivors and will be led by 2 trained therapists. Participants will complete four assessments (involving a clinician administered interview and standardized questions): pre-treatment, post- treatment, and 6 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of majority, with a history of breast cancer and who are at least 3 months following the end of their treatment
* Fluent in English
* Exceed the clinical cut-off for sexual distress (Female Sexual Distress Scale).
* Women who are, and who are not, in a relationship will be eligible as long as they have engaged in sexual activity either alone or with a sexual partner in the past 6 months, or as long as they indicate a willingness to engage in sexual activity (alone or with a sexual partner) during the time period of the study.

Exclusion Criteria:

* Active cancer treatment (e.g. chemotherapy or radiation, not including endocrine or maintenance therapies provided they remain constant for the study duration), or scheduled breast reconstruction during the study period.
* Borderline Personality Disorder or other psychiatric or medical conditions that preclude the ability to fully participate in the group sessions, assessments, and homework.
* In order to determine whether any changes in symptoms are a result of participation in the intervention, women must also agree to 1) not make changes to or commence vaginal interventions (e.g., topical hormone treatments, vaginal moisturizers, vaginal dilation) or 2) engage in other treatments for sexual difficulties (e.g., sex therapy), for 2 weeks prior to the baseline assessment until 2 weeks following the final intervention session.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
A Change from Baseline Sexual Interest and Desire Female (SIDI-F) Score at 2 weeks' post-treatment | Baseline/T1 is within 2 weeks pre-treatment and T2 is within 2 weeks post-treatment
  Sexual desire will be measured with the 13-item Sexual Interest and Desire Inventory which is a 14-item questionnaire that assesses sexual desire in women which includes one non-scored item assessing intercourse frequency. Possible total scores range from 0 - 51, with higher scores indicating higher levels of sexual functioning.
A Change from Baseline Sexual Interest and Desire Female (SIDI-F) Score at 6 month follow-up | Baseline/T1 is within 2 weeks pre-treatment and T3 is at 6 month follow-up
  Sexual desire will be measured with the 13-item Sexual Interest and Desire Inventory which is a 14-item questionnaire that assesses sexual desire in women which includes one non-scored item assessing intercourse frequency. Possible total scores range from 0 - 51, with higher scores indicating higher levels of sexual functioning.
No Change in Sexual Interest and Desire Female (SIDI-F) Score from 2 weeks' post-treatment (T2) and at 6 month follow-up (T3) | T2 is within 2 weeks post-treatment and T3 is at 6 month follow-up
  Sexual desire will be measured with the 13-item Sexual Interest and Desire Inventory which is a 14-item questionnaire that assesses sexual desire in women which includes one non-scored item assessing intercourse frequency. Possible total scores range from 0 - 51, with higher scores indicating higher levels of sexual functioning.
A Change from Baseline Female Sexual Distress Scale - Revised (FSDS-R) Score at 2 weeks' post-treatment | Baseline/T1 is within 2 weeks pre-treatment and T2 is within 2 weeks post-treatment
  Sexual distress will be assessed using the Female Sexual Distress Scale - Revised which is a 13-item scale where scores on the scale range from 0 - 52, where higher scores represent higher levels of distress.
A Change from Baseline Female Sexual Distress Scale - Revised (FSDS-R) Score at 6 month follow-up | Baseline/T1 is within 2 weeks pre-treatment and T3 is at 6 month follow-up
  Sexual distress will be assessed using the Female Sexual Distress Scale - Revised which is a 13-item scale where scores on the scale range from 0 - 52, where higher scores represent higher levels of distress.
No Change in Female Sexual Distress Scale - Revised (FSDS-R) Score from T2 at 2 weeks' post-treatment and at 6 month follow-up | T2 is within 2 weeks post-treatment and T3 is at 6 month follow-up
  Sexual distress will be assessed using the Female Sexual Distress Scale - Revised which is a 13-item scale where scores on the scale range from 0 - 52, where higher scores represent higher levels of distress.
A Change from Baseline Sexual Pain Rating Score at 2 weeks' post-treatment | Baseline/T1 is within 2 weeks pre-treatment and T2 is within 2 weeks post-treatment
  Numeric Rating Scale of 0-10 (from no pain to worst possible pain) in response to vaginal penetration.
A Change from Baseline Sexual Pain Rating Score at 6 month follow-up | Baseline/T1 is within 2 weeks pre-treatment and T3 is at 6 month follow-up
  Numeric Rating Scale of 0-10 (from no pain to worst possible pain) in response to vaginal penetration.
No Change in Sexual Pain Rating Score from 2 weeks' post-treatment and at 6 month follow-up | T2 is within 2 weeks post-treatment and T3 is at 6 month follow-up
  Numeric Rating Scale of 0-10 (from no pain to worst possible pain) in response to vaginal penetration.

CONTACTS AND LOCATIONS:
Locations (1):
- UBC Sexual Health Lab, Vancouver Hospital, Vancouver, British Columbia, Canada